CLINICAL TRIAL: NCT01419197
Title: A Phase III Randomized, Multicenter, Two Arm, Open-label Trial to Evaluate the Efficacy of Trastuzumab Emtansine Compared With Treatment of Physician's Choice in Patients With HER2-positive Metastatic Breast Cancer Who Have Received at Least Two Prior Regimens of HER2 Directed Therapy
Brief Title: A Study of Trastuzumab Emtansine in Comparison With Treatment of Physician's Choice in Participants With HER2-positive Breast Cancer Who Have Received at Least Two Prior Regimens of HER2-directed Therapy
Acronym: TH3RESA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TDM4997g; BO25734 (Other: Hoffmann-La Roche); 2011-000509-29 (EudraCT Number)
Record Dates: First submitted 2011-08-16; First posted 2011-08-18 (Estimated); Results first posted 2014-05-05 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Ado-Trastuzumab Emtansine

ARMS (2):
- Trastuzumab emtansine (Experimental): Trastuzumab emtansine 3.6 mg/kg intravenously every 3 weeks until disease progression (as assessed by the investigator) or unmanageable toxicity.
  Interventions: Drug: Trastuzumab emtansine
- Treatment of physician's choice (Active Comparator): Treatment of physician's choice until disease progression (as assessed by the investigator) or unmanageable toxicity. The treatments included single-agent chemotherapy, single-agent or dual-agent hormonal therapy for hormone receptor positive-disease, and HER2-directed therapy.
  Interventions: Drug: Treatment of physician's choice

INTERVENTIONS:
Drug: Trastuzumab emtansine — The dose was calculated based on the patient's Baseline weight on Day 1 of each 3-week treatment cycle. The same dose was administered in subsequent cycles if the patient's weight stayed within 10% of the Baseline weight. If there was a weight change > 10%, the dose was adjusted accordingly and the recorded weight became the new Baseline weight. Trastuzumab emtansine was provided as a single-use lyophilized formulation.
  Other Names: Kadcyla; T-DM1
  Arms: Trastuzumab emtansine
Drug: Treatment of physician's choice — The treatment of physician's choice (TPC) was a protocol-specified approved or standard of care therapy or combination of therapies, based on frequently used regimens for late-line HER2-positive metastatic breast cancer treatment after receipt of both trastuzumab- and lapatinib-containing regimens. The therapies included single-agent chemotherapy, single-agent (e.g., tamoxifen or aromatase inhibitor) or dual-agent (e.g., aromatase inhibitor with luteinizing hormone releasing hormone [LHRH] agonist) hormonal therapy for hormone receptor positive-disease, and HER2-directed therapy.
  Participants who had documented progressive disease (PD) were eligible to switch treatment to receive trastuzumab emtansine 3.6 mg/kg. Participants who switched treatment remained on trastuzumab emtansine treatment until another PD event or unmanageable toxicity.
  The formulation, storage, and preparation of all TPC were as per the appropriate package insert or national prescribing information.
  Arms: Treatment of physician's choice

SUMMARY:
This randomized, multicenter, 2-arm, open-label study (TH3RESA) will evaluate the efficacy and safety of trastuzumab emtansine (T-DM1) in comparison with treatment of the physician's choice in participants with metastatic or unresectable locally advanced/recurrent human epidermal growth factor receptor 2 (HER2)-positive breast cancer. Eligible participants will be randomized to receive either trastuzumab emtansine 3.6 mg/kg intravenously every 21 days or treatment of the physician's choice. Participants continue to receive study treatment until disease progression or unacceptable toxicity occurs. This study is also known under Roche study protocol number BO25734.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants ≥ 18 years of age.
* Histologically or cytologically documented breast cancer.
* Metastatic or unresectable locally advanced/recurrent breast cancer.
* HER2-positive disease by prospective laboratory confirmation.
* Disease progression on the last regimen received as defined by the investigator.
* Prior treatment with an trastuzumab, a taxane, and lapatinib.
* Disease progression after at least two regimens of HER2-directed therapy in the metastatic or unresectable locally advanced/recurrent setting.
* Adequate organ function, as evidenced by laboratory results.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Left ventricular ejection fraction (LVEF) ≥ 50% by echocardiogram or multi gated acquisition scan.

Exclusion Criteria:

* Chemotherapy ≤ 21 days before first study treatment.
* Trastuzumab ≤ 21 days before first study treatment.
* Lapatinib ≤ 14 days before first study treatment.
* Prior enrollment in a trastuzumab emtansine containing study, regardless whether the patient received prior trastuzumab emtansine.
* Brain metastases that are untreated or symptomatic, or require any radiation, surgery or corticosteroid therapy to control symptoms within 1 month of randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 602 (Actual)
Dates: Start 2011-09; Primary Completion 2013-02 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (166):
- United States (55):
  - Tucson, Arizona
  - Hot Springs, Arkansas
  - Hayward, California
  - Highland, California
  - Oakland, California
  - Roseville, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - San Jose, California
  - Santa Clara, California
  - South San Francisco, California
  - Stockton, California
  - Vallejo, California
  - Walnut Creek, California
  - West Hollywood, California
  - Denver, Colorado
  - Trumbull, Connecticut
  - Newark, Delaware
  - Washington D.C., District of Columbia
  - Coral Springs, Florida
  - Deerfield Beach, Florida
  - Fort Myers, Florida
  - Jacksonville, Florida
  - Plantation, Florida
  - Marietta, Georgia
  - Post Falls, Idaho
  - Chicago, Illinois
  - Maywood, Illinois
  - Fort Wayne, Indiana
  - Sioux City, Iowa
  - Wichita, Kansas
  - Scarborough, Maine
  - Bethesda, Maryland
  - Columbia, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Omaha, Nebraska
  - New Brunswick, New Jersey
  - Lake Success, New York
  - The Bronx, New York
  - Charlotte, North Carolina
  - Columbus, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Chattanooga, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - Fort Worth, Texas
  - San Antonio, Texas
  - Richmond, Virginia
  - Seattle, Washington
- Australia (4):
  - Kogarah, New South Wales
  - South Brisbane, Queensland
  - Frankston, Victoria
  - Perth, Western Australia
- Belgium (2):
  - Leuven
  - Wilrijk
- Brazil (6):
  - Salvador, Estado de Bahia
  - Goiânia, Goiás
  - Rio de Janeiro, Rio de Janeiro
  - Porto Alegre, Rio Grande do Sul
  - Itajaí, Santa Catarina
  - São Paulo, São Paulo
- Canada (5):
  - Moncton, New Brunswick
  - Toronto, Ontario
  - Québec, Quebec
  - Regina, Saskatchewan
  - Saskatoon, Saskatchewan
- Czechia (4):
  - Brno
  - Hradec Králové
  - Olomouc
  - Prague
- France (16):
  - Angers
  - Bordeaux
  - Caen
  - Lyon
  - Montpellier
  - Nantes
  - Nice
  - Nîmes
  - Paris
  - Reims
  - Rouen
  - Saint-Priest-en-Jarez
  - Strasbourg
  - Toulouse
  - Tours
  - Villejuif
- Germany (11):
  - Bielefeld
  - Hamburg
  - Hanover
  - Kiel
  - Mainz
  - München
  - Ravensburg
  - Recklinghausen
  - Stuttgart
  - Trier
  - Troisdorf
- Hungary (6):
  - Budapest
  - Gyula
  - Kecskemét
  - Miskolc
  - Szeged
  - Szolnok
- India (5):
  - Bangalore
  - Chennai
  - Kolkata
  - New Delhi
  - Pune
- Israel (7):
  - Beersheba
  - Hafia
  - Jerusalem
  - Petah Tikva
  - Ramat Gan
  - Rehovot
  - Tel Aviv
- Italy (8):
  - Potenza, Basilicate
  - Napoli, Campania
  - Genoa, Liguria
  - Bergamo, Lombardy
  - Brescia, Lombardy
  - Milan, Lombardy
  - Biella, Piedmont
  - Cona (Ferrara), Veneto
- Oslo, Norway
- Poland (6):
  - Bialystok
  - Bydgoszcz
  - Gdansk
  - Lublin
  - Poznan
  - Warsaw
- Russia (3):
  - Moscow
  - Samara
  - Stavropol
- Slovakia (2):
  - Košice
  - Poprad
- South Korea (2):
  - Kyunggi-do
  - Seoul
- Spain (8):
  - Barcelona, Barcelona
  - A Coruña, La Coruña
  - Madrid, Madrid
  - Málaga, Malaga
  - Murcia, Murcia
  - Seville, Sevilla
  - Valencia, Valencia
  - Bilbao, Vizcaya
- Sweden (3):
  - Örebro
  - Umeå
  - Uppsala
- Switzerland (2):
  - Bern
  - Zurich
- Bangkok, Thailand
- United Kingdom (9):
  - Brighton
  - Guildford
  - London
  - Maidstone
  - Metropolitan Borough of Wirral
  - Nottingham
  - Sheffield
  - Stoke-on-Trent
  - Westcliffe-on-sea

REFERENCES:
- [Derived] Chen SC, Quartino A, Polhamus D, Riggs M, French J, Wang X, Vadhavkar S, Smitt M, Hoersch S, Strasak A, Jin JY, Girish S, Li C. Population pharmacokinetics and exposure-response of trastuzumab emtansine in advanced breast cancer previously treated with >/=2 HER2-targeted regimens. Br J Clin Pharmacol. 2017 Dec;83(12):2767-2777. doi: 10.1111/bcp.13381. Epub 2017 Sep 3. PMID 28733983
- [Derived] Krop IE, Kim SB, Martin AG, LoRusso PM, Ferrero JM, Badovinac-Crnjevic T, Hoersch S, Smitt M, Wildiers H. Trastuzumab emtansine versus treatment of physician's choice in patients with previously treated HER2-positive metastatic breast cancer (TH3RESA): final overall survival results from a randomised open-label phase 3 trial. Lancet Oncol. 2017 Jun;18(6):743-754. doi: 10.1016/S1470-2045(17)30313-3. Epub 2017 May 16. PMID 28526538
- [Derived] Krop IE, Kim SB, Gonzalez-Martin A, LoRusso PM, Ferrero JM, Smitt M, Yu R, Leung AC, Wildiers H; TH3RESA study collaborators. Trastuzumab emtansine versus treatment of physician's choice for pretreated HER2-positive advanced breast cancer (TH3RESA): a randomised, open-label, phase 3 trial. Lancet Oncol. 2014 Jun;15(7):689-99. doi: 10.1016/S1470-2045(14)70178-0. Epub 2014 May 2. PMID 24793816

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 602 patients were randomized to the study (404 to receive Trastuzumab Emtansine and 198 to receive Treatment of Physician's Choice).
Groups:
- Treatment of Physician's Choice: Treatment of physician's choice until disease progression (as assessed by the investigator) or unmanageable toxicity. The treatments included single-agent chemotherapy, single-agent or dual-agent hormonal therapy for hormone receptor positive-disease, and human epidermal growth factor receptor 2 (HER2)-directed therapy.
Period: Overall Study
Arm/Group | Trastuzumab Emtansine | Treatment of Physician's Choice
Started | 404 | 198
Switched to Trastuzumab Emtansine | 0 | 94
Completed | 0 | 0
Not Completed | 404 | 198
Not completed — Death | 247 | 122
Not completed — Physician Decision | 4 | 4
Not completed — Non-compliance | 3 | 1
Not completed — Withdrawal by Subject | 33 | 32
Not completed — Study Completed by Sponsor | 103 | 34
Not completed — Reason Not Specified | 0 | 1
Not completed — Lost to Follow-up | 14 | 4

BASELINE CHARACTERISTICS:
Population: Randomized population: All participants who were randomized to the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Trastuzumab Emtansine | Treatment of Physician's Choice | Total
Number analyzed (Participants) | 404 | 198 | 602
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (10.4) | 54.3 (10.8) | 53.6 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 401 | 197 | 598
  Male | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the time from randomization to the first documented disease progression by investigator assessment using Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 or death from any cause, whichever occurred first. Progression-free survival was a co-primary endpoint.
Time Frame: Baseline to the clinical cut-off date of 11 Feb 2013 (up to 2 years)
Population: Randomized population: All participants who were randomized to the study. Participants were included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab Emtansine | Treatment of Physician's Choice
Number analyzed (Participants) | 404 | 198
Months | 6.2 [5.59 to 6.87] | 3.3 [2.89 to 4.14]
Statistical Analysis 1: Comparison: Trastuzumab Emtansine vs Treatment of Physician's Choice; The analysis was stratified for 1) World region (United States, Western Europe, or Other); 2) Number of prior regimens, excluding single-agent hormones, for treatment of metastatic or unresectable locally advanced/recurrent disease (≤ 3 or > 3); and 3) Presence of visceral disease (any visceral disease vs no visceral disease); Test type: Superiority or Other; p < 0.0001, Log Rank — The two-sided stratified log-rank test was used to compare progression-free survival between the two treatment arms at the overall two-sided significance level of 0.5%; Hazard Ratio (HR) = 0.528, 95% CI 2-sided [0.422 to 0.661] — The hazard ratio was estimated by Cox regression

2. Primary Outcome: Overall Survival
Description: Overall survival (OS) was defined as the time from randomization to death from any cause. Overall survival was a co-primary endpoint.
Time Frame: Baseline to the clinical cut-off date of 11 Feb 2013 (up to 2 years)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab Emtansine | Treatment of Physician's Choice
Number analyzed (Participants) | 404 | 198
Months | NA [13.14 to NA] — The median and the upper limit of the confidence interval could not be estimated due to too few events. | 14.9 [11.27 to NA] — The upper limit of the confidence interval could not be estimated due to too few events.
Statistical Analysis 1: Comparison: Trastuzumab Emtansine vs Treatment of Physician's Choice; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0034, Log Rank — The 2-sided stratified log-rank test was used at the overall two-sided significance level of 4.5%. The pre-specified O'Brien-Fleming stopping boundary for this first OS interim analysis was HR<0.363 (p-value < 0.0000013); Hazard Ratio (HR) = 0.552, 95% CI 2-sided [0.369 to 0.826] — The hazard ratio was estimated by Cox regression

3. Secondary Outcome: Percentage of Participants With an Objective Response
Description: An objective response was defined as a complete or partial response determined on 2 consecutive occasions ≥ 4 weeks apart using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Complete response was defined as the disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must be < 10 mm on the short axis. Partial response was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum. Participants who had no post-baseline tumor assessment were counted as non-responders.
Time Frame: Baseline to the clinical cut-off date of 11 Feb 2013 (up to 2 years)
Population: Randomized population: All participants who were randomized to the study. Only participants with measurable disease at Baseline were included in the analysis. Participants were included in the treatment group to which they were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trastuzumab Emtansine | Treatment of Physician's Choice
Number analyzed (Participants) | 345 | 163
Percentage of participants | 31.3 [26.5 to 36.5] | 8.6 [5.1 to 13.8]
Statistical Analysis 1: Comparison: Trastuzumab Emtansine vs Treatment of Physician's Choice; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mantel Haenszel; Difference in Response Percentage = 22.7, 95% CI 2-sided [16.2 to 29.2]

4. Secondary Outcome: Duration of the Objective Response
Description: Duration of the objective response was defined as the time from the first tumor assessment that was judged to indicate that the patient had an objective response to the time of first documented disease progression using RECIST v1.1 per investigator assessment or death from any cause, whichever occurred first.
Time Frame: Baseline to the clinical cut-off date of 11 Feb 2013 (up to 2 years)
Population: Randomized population: All participants who were randomized to the study. Only participants with an objective response were included in the analysis. Participants were included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab Emtansine | Treatment of Physician's Choice
Number analyzed (Participants) | 108 | 14
Months | 9.7 [6.60 to 10.51] | NA [2.40 to NA] — The median and the upper confidence interval value could not be estimated due to too few events.

5. Secondary Outcome: 6-month and 1-year Survival
Description: 6-month and 1-year survival were defined as the percentage of participants who were alive at 6 months and 1 year, respectively, as estimated using Kaplan-Meier method.
Time Frame: Baseline to the clinical cut-off date of 11 Feb 2013 (up to 2 years)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trastuzumab Emtansine | Treatment of Physician's Choice
Number analyzed (Participants) | 404 | 198
Percentage of participants
  6-Month Survival | 90.9 [87.79 to 94.01] | 78.3 [71.49 to 85.19]
  1-Year Survival | 68.6 [59.91 to 77.28] | 56.9 [42.22 to 71.63]
Statistical Analysis 1: Comparison: Trastuzumab Emtansine vs Treatment of Physician's Choice; 6-month survival; Test type: Superiority or Other; p = 0.0011, z-test — The p-value for the difference in survival rate was derived from the z-test using the standard errors computed using Greenwood's method; Difference in Survival Percentage = 12.6, 95% CI 2-sided [5.03 to 20.09]
Statistical Analysis 2: Comparison: Trastuzumab Emtansine vs Treatment of Physician's Choice; 1-year survival; Test type: Superiority or Other; p = 0.1805, z-test — The p-value for the difference in survival rates was derived from the z-test using the standard errors computed using Greenwood's method; Difference in Survival Percentage = 11.7, 95% CI 2-sided [-5.41 to 28.75]

6. Secondary Outcome: Time to Pain Symptom Progression
Description: Time to pain symptom progression was defined as the time from randomization to the first documentation of an increase in narcotic use and/or a 10 point increase from Baseline in the pain score as measured by the European Organisation for Research and Treatment of Cancer, Quality of Life Questionnaire for patients with bone metastases (EORTC QLQ-BM22). The EORTC QLQ-BM22 assesses the symptoms of bone metastases using 22 items: 5 items for sites of pain, 3 pain characteristics, 8 functional interference aspects, and 6 psychosocial aspects. The pain score was derived from the 3 pain characteristic items. Each item was rated on a 4-point scale, where 1=Not at all to 4=Very much. The pain score was the sum of the 3 pain characteristic scores and was normalized to a scale of 0 to 100. A higher score indicates greater pain.
Time Frame: Baseline to the clinical cut-off date of 11 Feb 2013 (up to 2 years)
Population: Randomized population: All participants who were randomized to the study. Only participants with a Baseline pain score and at least 1 post-baseline pain score were included in the analysis. Participants were included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab Emtansine | Treatment of Physician's Choice
Number analyzed (Participants) | 297 | 117
Months | 2.9 [2.2 to 3.7] | 3.6 [2.7 to 4.5]
Statistical Analysis 1: Comparison: Trastuzumab Emtansine vs Treatment of Physician's Choice; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4952, Log Rank; Hazard Ratio (HR) = 1.115, 95% CI 2-sided [0.819 to 1.517]

7. Secondary Outcome: Change From Baseline in the EORTC QLQ-BM22 Pain Score on Day 1 of Each Cycle
Description: The EORTC QLQ-BM22 assesses the symptoms of bone metastases using 22 items: 5 items for sites of pain, 3 pain characteristics, 8 functional interference aspects, and 6 psychosocial aspects. The pain score was derived from the 3 pain characteristic items. Each item was rated on a 4-point scale, where 1=Not at all to 4=Very much. The pain score was the sum of the 3 pain characteristic scores and was normalized to a scale of 0 to 100. A higher score indicates greater pain. A negative change score indicates improvement.
Time Frame: Baseline to the clinical cut-off date of 11 Feb 2013 (up to 2 years)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Trastuzumab Emtansine | Treatment of Physician's Choice
Number analyzed (Participants) | 297 | 117
Units on a scale
  Cycle 2 (n=282,98) | -3.4 (21.1) | -9.4 (22.1)
  Cycle 3 (n=257,86) | -4.6 (21.1) | -6.1 (21.4)
  Cycle 4 (n=236,74) | -4.8 (19.6) | -3.8 (24.1)
  Cycle 5 (n=224,54) | -6.6 (22.8) | -2.7 (18.9)
  Cycle 6 (n=195,42) | -4.8 (23.5) | 2.4 (17.1)
  Cycle 7 (n=163,30) | -4.2 (23.8) | -1.5 (15.6)
  Cycle 8 (n=130,20) | -7.0 (21.0) | 2.2 (18.6)
  Cycle 9 (n=97,15) | -5.8 (22.2) | 6.7 (20.1)
  Cycle 10 (n=80,7) | -8.9 (21.2) | 1.6 (11.9)
  Cycle 11 (n=56,8) | -10.5 (23.1) | 0.0 (8.4)
  Cycle 12 (n=48,7) | -11.3 (25.8) | 1.6 (7.7)
  Cycle 13 (n=40,5) | -10.0 (23.3) | 2.2 (12.2)
  Cycle 14 (n=33,5) | -10.1 (21.8) | 0.0 (7.9)
  Cycle 15 (n=27,3) | -13.2 (22.0) | 0.0 (0.0)
  Cycle 16 (n=19,3) | -12.3 (19.6) | -3.7 (6.4)
  Cycle 17 (n=15,2) | -7.4 (22.9) | -5.6 (7.9)
  Cycle 18 (n=11,0) | -9.1 (12.0) | NA (NA) — There were no participants with available data.
  Cycle 19 (n=8,0) | 1.4 (9.3) | NA (NA) — There were no participants with available data.
  Cycle 20 (n=4,0) | -5.6 (23.1) | NA (NA) — There were no participants with available data.
  Cycle 21 (n=3,0) | -3.7 (6.4) | NA (NA) — There were no participants with available data.
  Termination Visit (n=84,37) | -1.6 (21.8) | -9.0 (23.3)

8. Secondary Outcome: Overall Survival (Final Analysis)
Description: Overall survival was defined as the time from randomization to death from any cause.
Time Frame: Baseline to the clinical cut-off date of 13 Feb 2015 (up to 4 years)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab Emtansine | Treatment of Physician's Choice
Number analyzed (Participants) | 404 | 198
Months | 22.7 [19.35 to 27.47] | 15.8 [13.50 to 18.66]
Statistical Analysis 1: Comparison: Trastuzumab Emtansine vs Treatment of Physician's Choice; The analysis was stratified for 1) World region (United States, Western Europe, or Other); 2) Number of prior regimens, excluding single-agent hormones, for treatment of metastatic or unresectable locally advanced/recurrent disease (≤ 3 or > 3); and 3) Presence of visceral disease (any visceral disease versus no visceral disease); Test type: Superiority or Other; p = 0.0007, Log Rank — The two-sided stratified log-rank test was used at the overall two-sided significance level of 4.5%. The pre-specified O'Brien-Fleming stopping boundary for this second and final interim analysis was HR<0.748 (p value < 0.012); Hazard Ratio (HR) = 0.677, 95% CI 2-sided [0.539 to 0.850] — The hazard ratio was estimated by Cox regression

9. Secondary Outcome: 6-month and 1-year Survival (Final Analysis)
Description: as for outcome 5
Time Frame: Baseline to the clinical cut-off date of 13 Feb 2015 (up to 4 years)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trastuzumab Emtansine | Treatment of Physician's Choice
Number analyzed (Participants) | 404 | 198
Percentage of participants
  6-Month Survival | 91.3 [88.52 to 94.11] | 78.9 [72.78 to 85.04]
  1-Year Survival | 76.5 [72.23 to 80.79] | 65.6 [58.36 to 72.76]
Statistical Analysis 1: Comparison: Trastuzumab Emtansine vs Treatment of Physician's Choice; 6-month survival; Test type: Superiority or Other; p = 0.0003, z-test — [p-value comment as in outcome 5, analysis 1]; Difference in Survival Percentage = 12.4, 95% CI 2-sided [5.67 to 19.14]
Statistical Analysis 2: Comparison: Trastuzumab Emtansine vs Treatment of Physician's Choice; 1-year survival; Test type: Superiority or Other; p = 0.0104, z-test — [p-value comment as in outcome 5, analysis 2]; Difference in Survival Percentage = 11.0, 95% CI 2-sided [2.58 to 19.33]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from treatment initiation until 30 days following the last administration of study drug or study discontinuation on 31 August 2015 (up to approximately 4 years).
Description: Safety population: All participants who received any amount of planned study treatment, according to treatment actually received. Data for participants in the Treatment of Physicians Choice (TPC) arm who switched treatment to receive trastuzumab emtansine (TE) following disease progression on TPC are presented separately. Median treatment duration of trastuzumab emtansine: 5.2 months (range 0.03-40.7),TPC: 2.7 months (range 0.03-31.0) and TE - Post TPC Treatment Switch: 4.5 months (range 1-43).
Groups:
- Treatment of Physician's Choice (TPC): Treatment of physician's choice until disease progression (as assessed by the investigator) or unmanageable toxicity. The treatments included single-agent chemotherapy, single-agent or dual-agent hormonal therapy for hormone receptor positive-disease, and HER2-directed therapy.
- Trastuzumab Emtansine - Post TPC Treatment Switch: Participants, who switched treatment in the Treatment of Physician's Choice arm to trastuzumab emtansine, were administered trastuzumab emtansine 3.6 mg/kg intravenously every 3 weeks until disease progression (as assessed by the investigator) or unmanageable toxicity.
Arm/Group | Trastuzumab Emtansine | Treatment of Physician's Choice (TPC) | Trastuzumab Emtansine - Post TPC Treatment Switch
Serious Adverse Events (participants affected / at risk) | 102/403 | 41/184 | 19/94
Other Adverse Events (participants affected / at risk) | 371/403 | 148/184 | 74/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab Emtansine (N=403) | Treatment of Physician's Choice (TPC) (N=184) | Trastuzumab Emtansine - Post TPC Treatment Switch (N=94)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 7 | 0
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Hypercalcaemia of malignancy (Endocrine disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0
Obstruction gastric (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Proctitis Haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 2 | 0
Adverse drug reaction (General disorders) | 1 | 0 | 0
Asthenia (General disorders) | 3 | 0 | 0
Death (General disorders) | 1 | 0 | 0
Device occlusion (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 2 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 2 | 2 | 0
Pain (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 7 | 2 | 1
Vessel puncture site haemorrhage (General disorders) | 1 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Nodular regenerative hyperplasia (Hepatobiliary disorders) | 3 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 4 | 1
Clostridium bacteraemia (Infections and infestations) | 0 | 1 | 0
Device related infection (Infections and infestations) | 1 | 1 | 0
Device related sepsis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 0
Infected fistula (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 2 | 0 | 0
Infectious colitis (Infections and infestations) | 0 | 1 | 0
Lung infection (Infections and infestations) | 1 | 0 | 1
Lymphangitis (Infections and infestations) | 1 | 0 | 0
Mastitis (Infections and infestations) | 0 | 1 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 1 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 5 | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 3 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 0
Tracheitis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 4 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 0 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound decomposition (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 | 1 | 0
Transaminases increased (Investigations) | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 0 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ataxia (Nervous system disorders) | 1 | 1 | 0
Brain oedema (Nervous system disorders) | 1 | 0 | 0
Cerebral haematoma (Nervous system disorders) | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 2 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Paraparesis (Nervous system disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 5 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Visual field defect (Nervous system disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Non-cardiogenic pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 0
Embolism (Vascular disorders) | 1 | 0 | 0
Embolism venous (Vascular disorders) | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 1 | 1
Superior vena cava syndrome (Vascular disorders) | 1 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 1
Abdominal infection (Infections and infestations) | 0 | 0 | 1
Abscess (Infections and infestations) | 0 | 0 | 1
Biliary tract infection (Infections and infestations) | 0 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 1
Hemiplegia (Nervous system disorders) | 0 | 0 | 1
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab Emtansine (N=403) | Treatment of Physician's Choice (TPC) (N=184) | Trastuzumab Emtansine - Post TPC Treatment Switch (N=94)
Anaemia (Blood and lymphatic system disorders) | 45 | 19 | 7
Leukopenia (Blood and lymphatic system disorders) | 9 | 11 | 0
Neutropenia (Blood and lymphatic system disorders) | 30 | 39 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 81 | 6 | 17
Abdominal pain (Gastrointestinal disorders) | 27 | 20 | 9
Constipation (Gastrointestinal disorders) | 90 | 32 | 7
Diarrhoea (Gastrointestinal disorders) | 52 | 40 | 10
Dry mouth (Gastrointestinal disorders) | 51 | 2 | 9
Dyspepsia (Gastrointestinal disorders) | 21 | 12 | 0
Gingival bleeding (Gastrointestinal disorders) | 21 | 0 | 0
Nausea (Gastrointestinal disorders) | 144 | 40 | 16
Stomatitis (Gastrointestinal disorders) | 13 | 11 | 0
Vomiting (Gastrointestinal disorders) | 77 | 16 | 10
Asthenia (General disorders) | 76 | 33 | 15
Chills (General disorders) | 21 | 4 | 0
Fatigue (General disorders) | 123 | 48 | 10
Influenza like illness (General disorders) | 21 | 2 | 0
Mucosal inflammation (General disorders) | 17 | 10 | 7
Oedema peripheral (General disorders) | 26 | 11 | 0
Pyrexia (General disorders) | 77 | 22 | 14
Nasopharyngitis (Infections and infestations) | 35 | 12 | 6
Upper respiratory tract infection (Infections and infestations) | 35 | 8 | 8
Urinary tract infection (Infections and infestations) | 26 | 7 | 9
Alanine aminotransferase increased (Investigations) | 38 | 10 | 7
Aspartate aminotransferase increased (Investigations) | 51 | 13 | 13
Blood alkaline phosphatase increased (Investigations) | 21 | 5 | 7
Blood bilirubin increased (Investigations) | 38 | 2 | 5
Ejection fraction decreased (Investigations) | 11 | 12 | 0
Decreased appetite (Metabolism and nutrition disorders) | 66 | 25 | 15
Hypokalaemia (Metabolism and nutrition disorders) | 30 | 4 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 60 | 8 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 35 | 13 | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 22 | 7 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 26 | 9 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 18 | 10 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 47 | 14 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 44 | 9 | 0
Dizziness (Nervous system disorders) | 31 | 6 | 6
Headache (Nervous system disorders) | 100 | 22 | 16
Neuropathy peripheral (Nervous system disorders) | 20 | 10 | 7
Paraesthesia (Nervous system disorders) | 28 | 11 | 9
Insomnia (Psychiatric disorders) | 35 | 6 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 76 | 24 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 42 | 21 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 67 | 7 | 12
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 20 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 23 | 17 | 0
Rash (Skin and subcutaneous tissue disorders) | 27 | 19 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 5
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 7
Pain (General disorders) | 0 | 0 | 5
Sinusitis (Infections and infestations) | 0 | 0 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.